CLINICAL TRIAL: NCT01414153
Title: Phase 2a, Multicenter, Masked, Randomized, Comparator Controlled Study Evaluating iSONEP™ as Monotherapy or Adjunctive Therapy to Lucentis/Avastin/Eylea Versus Lucentis/Avastin/Eylea Alone for Treatment of Subjects With Choroidal Neovascularization (CNV) Secondary to Age-related Macular Degeneration (AMD)
Brief Title: Efficacy and Safety Study of iSONEP With & Without Lucentis/Avastin/Eylea to Treat Wet AMD
Acronym: Nexus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lpath, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LT1009-Oph-003
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Results first posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-08

CONDITIONS: Exudative Age-related Macular Degeneration
Keywords: choroidal neovascularization; age-related macular degeneration; iSONEP; sonepcizumab; Lucentis; ranibizumab; Avastin; bevacizumab; Eylea; aflibercept
MeSH Terms: conditions — Choroidal Neovascularization; Macular Degeneration | interventions — sonepcizumab; Ranibizumab; Bevacizumab; aflibercept; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Monotherapy (Experimental): 4.0 mg iSONEP followed by sham injection; given monthly intravitreously for 4 months
  Interventions: Drug: 4.0 mg iSONEP; Drug: sham injection
- 0.5 mg iSONEP & Lucentis/Avastin/Eylea (Experimental): 0.5 mg iSONEP and 0.5 mg Lucentis or 1.25 mg Avastin or 2 mg Eylea; given monthly intravitreously for 4 months
  Interventions: Drug: 0.5 mg iSONEP; Drug: 0.5 mg Lucentis or 1.25 mg Avastin or 2 mg Eylea
- 4.0 mg iSONEP & Lucentis/Avastin/Eylea (Experimental): 4.0 mg iSONEP followed by 0.5 mg Lucentis or 1.25 mg Avastin or 2 mg Eylea; given monthly intravitreously for 4 months
  Interventions: Drug: 4.0 mg iSONEP; Drug: 0.5 mg Lucentis or 1.25 mg Avastin or 2 mg Eylea
- Lucentis or Avastin or Eylea (Active Comparator): 0.5 mg Lucentis or 1.25 mg Avastin or 2 mg Eylea followed by a sham injection; given monthly intravitreously for 4 months
  Interventions: Drug: 0.5 mg Lucentis or 1.25 mg Avastin or 2 mg Eylea; Drug: sham injection

INTERVENTIONS:
Drug: 4.0 mg iSONEP — 4.0 mg iSONEP given monthly intravitreously for 4 months
  Other Names: sonepcizumab
  Arms: 4.0 mg iSONEP & Lucentis/Avastin/Eylea; Monotherapy
Drug: 0.5 mg iSONEP — 0.5 mg iSONEP given monthly intravitreously for 4 months
  Other Names: sonepcizumab
  Arms: 0.5 mg iSONEP & Lucentis/Avastin/Eylea
Drug: 0.5 mg Lucentis or 1.25 mg Avastin or 2 mg Eylea — 0.5 mg Lucentis or 1.25 mg Avastin or 2 mg Eylea given monthly intravitreously for 4 months
  Other Names: ranibizumab; bevacizumab; aflibercept
  Arms: 0.5 mg iSONEP & Lucentis/Avastin/Eylea; 4.0 mg iSONEP & Lucentis/Avastin/Eylea; Lucentis or Avastin or Eylea
Drug: sham injection — administered monthly for 4 months
  Other Names: placebo
  Arms: Lucentis or Avastin or Eylea; Monotherapy

SUMMARY:
The purpose of the study is to determine the safety and efficacy of 4 monthly injections of iSONEP given alone or in combination with Lucentis, Avastin or Eylea in subjects with wet Age-related Macular Degeneration (AMD). iSONEP not only has an anti-permeability effect, but also has anti-angiogenic, anti-inflammatory, and anti-fibrotic properties. The drug may therefore have the ability to achieve better visual outcomes than Lucentis, Avastin or Eylea, particularly in those subjects who do not demonstrate a robust response to Lucentis, Avastin or Eylea after several monthly injections. Further, the combination of Lucentis, Avastin or Eylea and iSONEP may be additive or synergistic. By inhibiting the multiple mechanisms that contribute to exudative-AMD-related vision loss, better visual outcomes may be possible than with Lucentis, Avastin or Eylea alone.

DETAILED DESCRIPTION:
The study will be conducted in subjects who qualify as "sub-responders" to Lucentis, Avastin or Eylea meaning that each subject has (i) residual subretinal or intra-retinal fluid observed on Cirrus or Spectralis Spectral Domain Optical Coherence Tomography (SD-OCT), (ii) leakage on fluorescein angiogram (FA), and (iii) an average central subfield thickness of ≥250 μm. Additionally, each subject will have previously received a minimum of 3 intravitreous (IVT) injections of Lucentis, Avastin or Eylea within the 12-month period prior to screening. Screening must occur between 28 and 65 days from the subject's last Lucentis or Avastin treatment or between 42 and 79 days from the subject's last Eylea treatment. Subjects must be dosed within 14 days of screening, and as of the day of initial study treatment (Day 0), meet the following criteria: (i) Early Treatment Diabetic Retinopathy Study (ETDRS) Best-corrected visual acuity (BCVA) of ≥25 and ≤73 letters (approximately 20/320 and 20/40 on the Snellen scale), (ii) residual subretinal or intra-retinal fluid observed on Cirrus or Spectralis SDOCT, and (iii) leakage on FA.

ELIGIBILITY:
Inclusion Criteria:

* ≥50 years of age with a diagnosis of wet AMD
* Subjects who have received 3 injections of Lucentis or Avastin or Eylea within 12 months prior to screening
* Active subfoveal CNV secondary to AMD (leakage on FA)
* Presence of residual subretinal or intraretinal fluid on Cirrus or Spectralis SDOCT
* SDOCT in the 1 mm central macular subfield on the retinal map analysis of ≥250 μm at screening
* ETDRS BCVA of ≥25 and ≤73 letters (approximately 20/320 and 20/40 on the Snellen scale) at screening and on Day 0
* In the fellow eye, ETDRS BCVA of 20/400 or better
* Subject with serous pigment epithelial detachment (PED) (any part of which may be subfoveal) with intraretinal and/or subretinal fluid may be included

Exclusion Criteria:

* Most recent IVT injection of Lucentis or Avastin fewer than 28 days and more than 65 days prior to screening
* Most recent IVT injection of Eylea fewer than 42 days and more than 79 days prior to screening
* Previous photodynamic therapy (PDT) or Macugen® at any time point
* Focal thermal laser or grid laser within 3 months prior to Day 0
* Use of IVT, subtenon or subconjunctival steroids within 3 months prior to Day 0
* Use of topical ophthalmic corticosteroids 2 weeks prior to Day 0
* Intraocular surgery, including cataract surgery, and / or laser of any type within 3 months prior to Day 0 or anticipated need for ocular surgery or ophthalmic laser treatment during the study period
* Subjects previously treated with, or are currently receiving treatment with another investigational agent or device for neovascular AMD in the study eye
* Retinal total lesion size >12 disc areas (30.5 mm2), including blood, scars and neovascularization as assessed by FA in the study eye
* Presence of a fibrovascular PED extending underneath the center of the fovea
* Presence of retinal angiomatous proliferation (RAP) lesions
* Presence of polypoidal choroidal vasculopathy (PCV) (if suspected, Indocyanine Green Angiography (ICG) should be performed at the discretion of the Investigator)
* Subretinal hemorrhage in the study eye if any of the following is true: (i) the subretinal hemorrhage represents 50% or more of the total lesion area; (ii) subfoveal blood is 1 or more disc areas in size (iii) subfoveal blood where the fovea is surrounded by less than 270 degrees of visible CNV on FA
* Scar or fibrosis making up >50% of total lesion area in the study eye
* Anatomic damage to the center of the fovea including fibrosis, scarring or atrophy
* History of a retinal pigment epithelial tear
* History of vitreous hemorrhage within 4 weeks prior to screening in the study eye
* Clinical evidence of diabetic retinopathy, diabetic macular edema or any other vascular disease affecting the retina, other than AMD, in either eye
* Uncontrolled glaucoma defined as: (i) as intraocular pressure ≥25 mmHg despite treatment with anti glaucoma medication in the study eye or (ii) by the Investigator
* Prior trabeculectomy or other filtration surgery in the study eye (prior laser trabeculoplasty is allowed)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2012-08; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dario A Paggiarino, MD, Study Director — Lpath, Inc.
Locations (44):
- United States (44):
  - Retina Consultants of Arizona, Peoria, Arizona
  - Retina Consultants of Arizona, Phoenix, Arizona
  - Associated Retina Consultants, Phoenix, Arizona
  - Retina Centers, P.C., Tucson, Arizona
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Retinal Diagnostic Center, Campbell, California
  - Specialty Eye Care Medical Center, Glendale, California
  - Retina Associates of Orange County, Laguna Hills, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Sagar Kenyon American Eye Institute, New Albany, California
  - Retinal Consultants Medical Group, Inc., Sacramento, California
  - Orange County Retina Medical Group, Santa Ana, California
  - Miramar Eye Specialists, Ventura, California
  - Florida Eye Microsurgical Institute, Boynton Beach, Florida
  - Retina Health Center, Fort Myers, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - East Florida Eye Institute, Stuart, Florida
  - Center for Retina & Macular Disease, Winter Haven, Florida
  - Retina Consultants of Hawaii, ‘Aiea, Hawaii
  - Midwest Eye Institute, Indianapolis, Indiana
  - Central Plains Eye MDs, Wichita, Kansas
  - Bennett & Bloom Eye Centers, Louisville, Kentucky
  - Retina Group of Washington, Chevy Chase, Maryland
  - Retina Specialists, Towson, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - TLC Eye Care and Laser Center, Jackson, Michigan
  - Retina Consultants of Michigan, Southfield, Michigan
  - Island Retina, Shirley, New York
  - Charlotte Eye Ear Nose & Throat Associates, Charlotte, North Carolina
  - Retina & Vitreous Center SO, Ashland, Oregon
  - Associates in Ophthalmology, West Mifflin, Pennsylvania
  - Palmetto Retina Center, West Columbia, South Carolina
  - Retina Research Institute of Texas, Abilene, Texas
  - Austin Retina Associates, Austin, Texas
  - Retina Research Center, Austin, Texas
  - Texas Retina Associates, Dallas, Texas
  - Valley Retina Institute, Harlingen, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retina Associates of South Texas, San Antonio, Texas
  - Rocky Mountain Retina Consultants, Salt Lake City, Utah
  - Retina Group of Washington, Fairfax, Virginia
  - Spokane Eye Clinical Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Monotherapy | 0.5 mg iSONEP & Lucentis/Avastin/Eylea | 4.0 mg iSONEP & Lucentis/Avastin/Eylea | Lucentis or Avastin or Eylea
Started | 38 | 40 | 39 | 41
Completed | 30 | 38 | 35 | 37
Not Completed | 8 | 2 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Monotherapy | 0.5 mg iSONEP & Lucentis/Avastin/Eylea | 4.0 mg iSONEP & Lucentis/Avastin/Eylea | Lucentis or Avastin or Eylea | Total
Number analyzed (Participants) | 38 | 40 | 39 | 41 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.1 (7.53) | 77.2 (7.43) | 77.6 (7.86) | 76.5 (7.95) | 76.8 (7.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 21 | 20 | 83
  Male | 16 | 20 | 18 | 21 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 2 | 3 | 10
  Not Hispanic or Latino | 36 | 37 | 37 | 38 | 148
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 0 | 2
  White | 36 | 39 | 39 | 40 | 154
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 38 | 40 | 39 | 41 | 158
Best Corrected Visual Acuity (ETDRS) [Mean (Standard Deviation); unit: letters] — Visual function was assessed using the ETDRS protocol, for which numerical scores range from 0 to 100 (roughly equivalent to 20/10 vision as measured by Snellen). A higher score (more letters read) represents better functioning.
  letters | 56.2 (15.84) | 58.7 (10.75) | 61.3 (9.20) | 63.2 (7.88) | 59 (11.45)
Choroidal neovascularization (CNV) Lesion Type [Number; unit: percentage of participants]
  Predominantly Classic | 10.5 | 15.0 | 12.8 | 22.0 | 60.3
  Minimally Classic | 5.3 | 5.0 | 5.1 | 7.3 | 22.7
  Occult | 76.3 | 77.5 | 79.5 | 61.0 | 294.3
  Unreadable | 5.3 | 0.0 | 0.0 | 2.4 | 7.7
  Missing | 2.6 | 2.5 | 2.6 | 7.3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Best Corrected Visual Acuity (BCVA) by Early Treatment Diabetic Retinopathy Study (ETDRS)
Description: Visual function was assessed using the ETDRS protocol, for which numerical scores range from 0 to 100 (roughly equivalent to 20/10 vision as measured by Snellen). A higher score represents better functioning. A positive number represents an increase in number of letters read correctly.
Time Frame: Baseline to Day 120
Population: Intent-to-treat (ITT) Population
Measure: Least Squares Mean (Standard Deviation); unit: letters
Arm/Group | Monotherapy | 0.5 mg iSONEP & Lucentis/Avastin/Eylea | 4.0 mg iSONEP & Lucentis/Avastin/Eylea | Lucentis or Avastin or Eylea
Number analyzed (Participants) | 38 | 40 | 39 | 41
letters | -3.17 (1.515) | 4.22 (1.459) | 3.63 (1.478) | 4.34 (1.455)

2. Secondary Outcome: Mean Change in Central Subfield Retinal Thickness
Time Frame: Baseline to Day 120
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: μM
Arm/Group | Monotherapy | 0.5 mg iSONEP & Lucentis/Avastin/Eylea | 4.0 mg iSONEP & Lucentis/Avastin/Eylea | Lucentis or Avastin or Eylea
Number analyzed (Participants) | 38 | 40 | 39 | 40
μM | 12.9 (12.45) | -72.4 (12.06) | -46.9 (12.20) | -67.7 (12.07)

3. Secondary Outcome: Mean Change in CNV Lesion Area as Determined by Fluorescein Angiography (FA).
Time Frame: Baseline to Day 120
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: mm^2
Arm/Group | Monotherapy | 0.5 mg iSONEP & Lucentis/Avastin/Eylea | 4.0 mg iSONEP & Lucentis/Avastin/Eylea | Lucentis or Avastin or Eylea
Number analyzed (Participants) | 30 | 40 | 39 | 40
mm^2 | 0.02 (0.793) | -4.91 (0.765) | -4.71 (0.775) | -5.30 (0.762)

4. Secondary Outcome: Proportion of Subjects Gaining Greater Than or Equal to 0, 5, 10 and 15 Letters on the ETDRS Chart.
Description: as for outcome 1
Time Frame: Baseline to Day 120
Measure: Number (80% Confidence Interval); unit: percentage of subjects
Arm/Group | Monotherapy | 0.5 mg iSONEP & Lucentis/Avastin/Eylea | 4.0 mg iSONEP & Lucentis/Avastin/Eylea | Lucentis or Avastin or Eylea
Number analyzed (Participants) | 38 | 40 | 39 | 41
percentage of subjects
  ≥ 0 letters gained | 44.7 [33.5 to 56.4] | 72.5 [61.5 to 81.7] | 71.8 [60.6 to 81.2] | 80.5 [70.2 to 88.3]
  ≥ 5 letters gained | 23.7 [14.8 to 34.8] | 42.5 [31.7 to 53.9] | 46.2 [35.0 to 57.6] | 53.7 [42.5 to 64.5]
  ≥ 10 letters gained | 13.2 [6.5 to 23.0] | 22.5 [14.1 to 33.2] | 28.2 [18.8 to 39.4] | 22.0 [13.7 to 32.4]
  ≥ 15 letters gained | 5.3 [1.4 to 13.4] | 15.0 [8.1 to 24.8] | 5.1 [1.4 to 13.1] | 0 [0.0 to 5.5]

5. Secondary Outcome: Proportion of Subjects Losing 3 Lines or More in ETDRS BCVA.
Description: Visual function was assessed using the ETDRS protocol, for which numerical scores range from 0 to 100 (roughly equivalent to 20/10 vision as measured by Snellen). A higher score represents better functioning. A positive number represents an increase in number of letters read correctly. One line is equivalent to 5 letters, so a loss of 3 lines is a loss of 15 letters.
Time Frame: Baseline to Day 120
Measure: Number (80% Confidence Interval); unit: percentage of subjects
Arm/Group | Monotherapy | 0.5 mg iSONEP & Lucentis/Avastin/Eylea | 4.0 mg iSONEP & Lucentis/Avastin/Eylea | Lucentis or Avastin or Eylea
Number analyzed (Participants) | 38 | 40 | 39 | 41
percentage of subjects
  ≥ 1 letters lost | 55.3 [43.6 to 66.5] | 27.5 [18.3 to 38.5] | 28.2 [18.8 to 39.4] | 19.5 [11.7 to 29.8]
  ≥ 5 letters lost | 44.7 [33.5 to 56.4] | 12.5 [6.2 to 22.0] | 17.9 [10.3 to 28.3] | 7.3 [2.7 to 15.6]
  ≥ 10 letters lost | 18.4 [10.6 to 29.0] | 7.5 [2.8 to 15.9] | 10.3 [4.5 to 19.5] | 2.4 [0.3 to 9.2]
  ≥ 15 letters lost | 10.5 [4.7 to 19.9] | 2.5 [0.3 to 9.4] | 5.1 [1.4 to 13.1] | 0.0 [0.0 to 5.5]

6. Secondary Outcome: Proportion of Subjects With ETDRS BCVA of 20/40 or Better.
Description: Visual function was assessed using the ETDRS protocol, for which numerical scores range from 0 to 100 (roughly equivalent to 20/10 vision as measured by Snellen). A higher score represents better functioning. A positive number represents an increase in number of letters read correctly. 20/40 Snellen corresponds to a range of 69-73 letters by ETDRS.
Time Frame: Baseline to Day 120
Measure: Number (80% Confidence Interval); unit: percentage of subjects
Arm/Group | Monotherapy | 0.5 mg iSONEP & Lucentis/Avastin/Eylea | 4.0 mg iSONEP & Lucentis/Avastin/Eylea | Lucentis or Avastin or Eylea
Number analyzed (Participants) | 38 | 40 | 39 | 41
percentage of subjects | 26.3 [17.0 to 37.6] | 47.5 [36.4 to 58.8] | 41 [30.2 to 52.6] | 56.1 [44.9 to 66.8]

7. Secondary Outcome: Proportion of Subjects With Adverse Events.
Time Frame: Baseline to Day 120
Measure: Number; unit: percentage of subjects
Arm/Group | Monotherapy | 0.5 mg iSONEP & Lucentis/Avastin/Eylea | 4.0 mg iSONEP & Lucentis/Avastin/Eylea | Lucentis or Avastin or Eylea
Number analyzed (Participants) | 38 | 40 | 39 | 41
percentage of subjects | 81.6 | 80.0 | 82.1 | 75.6

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of consent through the last study visit.
Description: Adverse events presented here are those that were treatment-emergent (those with an onset date on or after the time of first dose).
Arm/Group | Monotherapy | 0.5 mg iSONEP & Lucentis/Avastin/Eylea | 4.0 mg iSONEP & Lucentis/Avastin/Eylea | Lucentis or Avastin or Eylea
Serious Adverse Events (participants affected / at risk) | 6/38 | 4/40 | 4/39 | 6/41
Other Adverse Events (participants affected / at risk) | 31/38 | 32/40 | 32/39 | 31/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy (N=38) | 0.5 mg iSONEP & Lucentis/Avastin/Eylea (N=40) | 4.0 mg iSONEP & Lucentis/Avastin/Eylea (N=39) | Lucentis or Avastin or Eylea (N=41)
angina unstable (Cardiac disorders) | 0 | 0 | 0 | 3
cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 1
coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0
myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
sick sinus syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
optic ischaemic neuropathy (Eye disorders) | 1 | 0 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
upper gastrointestinal bleed (Gastrointestinal disorders) | 0 | 1 | 0 | 0
chest pain (General disorders) | 1 | 0 | 0 | 1
anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1
pneumonia (Infections and infestations) | 0 | 0 | 2 | 1
pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 1
hypotension (Vascular disorders) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy (N=38) | 0.5 mg iSONEP & Lucentis/Avastin/Eylea (N=40) | 4.0 mg iSONEP & Lucentis/Avastin/Eylea (N=39) | Lucentis or Avastin or Eylea (N=41)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0
Corneal dystrophy (Congenital, familial and genetic disorders) | 0 | 0 | 2 | 2
Age-related macular degeneration (Eye disorders) | 2 | 0 | 0 | 0
Anterior chamber cell (Eye disorders) | 1 | 3 | 0 | 2
Anterior chamber flare (Eye disorders) | 0 | 1 | 2 | 2
Cataract nuclear (Eye disorders) | 0 | 3 | 0 | 0
Cataract subcapsular (Eye disorders) | 0 | 2 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 13 | 24 | 21 | 17
Corneal oedema (Eye disorders) | 0 | 0 | 2 | 2
Eye haemorrhage (Eye disorders) | 0 | 0 | 2 | 0
Eye irritation (Eye disorders) | 0 | 2 | 1 | 2
Eye pain (Eye disorders) | 2 | 3 | 6 | 3
Eye pruritus (Eye disorders) | 1 | 2 | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 2 | 0 | 0
Macular degeneration (Eye disorders) | 2 | 0 | 1 | 0
Punctate keratitis (Eye disorders) | 2 | 0 | 1 | 0
Retinal haemorrhage (Eye disorders) | 11 | 0 | 3 | 1
Visual acuity reduced (Eye disorders) | 1 | 1 | 2 | 1
Vitreous detachment (Eye disorders) | 2 | 3 | 1 | 3
Vitreous floaters (Eye disorders) | 3 | 5 | 8 | 5
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 3 | 1
Cystitis (Infections and infestations) | 0 | 4 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 3 | 0 | 3
Pneumonia (Infections and infestations) | 0 | 1 | 2 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 3 | 1
Urinary tract infection (Infections and infestations) | 2 | 3 | 2 | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 4
Activated partial thromboplastin time prolonged (Investigations) | 1 | 5 | 0 | 2
Intraocular pressure increased (Investigations) | 0 | 1 | 11 | 2
Prothrombin time prolonged (Investigations) | 0 | 1 | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 2 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | 1
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3
Hypertension (Vascular disorders) | 1 | 2 | 3 | 2
Hypotension (Vascular disorders) | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days